CLINICAL TRIAL: NCT03768817
Title: A Retrospective Chart Review Study to Assess the Clinical Outcome of Triheptanoin Treatment in Patients With Long-chain Fatty Acid Oxidation Disorders (LC-FAOD) Treated Under Expanded Access Program
Brief Title: Clinical Outcome of Triheptanoin Treatment in Patients With Long-chain Fatty Acid Oxidation Disorders (LC-FAOD) Treated Under Expanded Access Program
Status: Completed | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX007-CL003
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Long-chain Fatty Acid Oxidation Disorders (LC-FAOD)
Keywords: Long-chain Fatty Acid Oxidation Disorders (LC-FAOD); Triheptanoin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with triheptanoin: Patients with LC-FAOD treated with triheptanoin before 01 September 2018 under eIND
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional retrospective medical record review study. No study investigational product will be administered in this protocol.

SUMMARY:
The primary objective of the study is to evaluate the clinical outcomes for the trigger event of patients who receive triheptanoin in the emergency Investigational New Drug (eIND) program.

DETAILED DESCRIPTION:
The study is a retrospective chart review of patients in the USA with LC-FAOD who received triheptanoin via eIND request from their metabolic or treating physician before 01 September 2018. Participating study sites will provide the medical records of subjects who meet eligibility criteria, and relevant data regarding the trigger event (the reason the patient was placed on triheptanoin) and key details about hospitalizations during the study period will be extracted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of any age with confirmed diagnosis of one of the LC-FAOD disorders including: mitochondrial trifunctional protein (TFP) deficiency, carnitine palmitoyltransferase deficiencies (CPT I and CPT II), very long chain acyl-CoA dehydrogenase (VLCAD) deficiency, long-chain 3-hydroxy-acyl-CoA dehydrogenase (LCHAD) deficiency, and carnitine acylcarnitine translocase (CATR) deficiency
* Treatment initiation with triheptanoin was via eIND before 01 September 2018
* Treated with triheptanoin in the USA
* Willing and able to provide written, signed informed consent, or where appropriate for subjects under the age of 18, or provide written assent and written informed consent by a legally authorized representative after the nature of the study has been explained and prior to any research-related procedures. To obtain and review medical records of deceased individuals, informed consent from next of kin or appropriate legal entity will be obtained, as applicable.

Exclusion Criteria:

* Unwilling to sign informed consent or assent to release of medical records

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Medical records of patients in the USA with LC-FAOD who received triheptanoin via eIND request from their metabolic or treating physician before 01 September 2018.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Duration of Hospitalization for Trigger Event | Up to 48 Weeks Prior to and 48 Weeks After the Start of Triheptanoin Treatment
Disposition on Discharge of Trigger Event | Up to 48 Weeks Prior to and 48 Weeks After the Start of Triheptanoin Treatment
Duration of Important Interventions for Trigger Event | Up to 48 Weeks Prior to and 48 Weeks After the Start of Triheptanoin Treatment
Number of Critical Medical Assessments Related to LC-FAOD for Trigger Event | Up to 48 Weeks Prior to and 48 Weeks After the Start of Triheptanoin Treatment

SECONDARY OUTCOMES:
Duration of Hospitalization for Other Major Clinical Events | Up to 48 Weeks Prior to and 48 Weeks After the Start of Triheptanoin Treatment
Disposition on Discharge of Other Major Clinical Events | Up to 48 Weeks Prior to and 48 Weeks After the Start of Triheptanoin Treatment
Number of Important Medical Interventions for Other Major Clinical Events | Up to 48 Weeks Prior to and 48 Weeks After the Start of Triheptanoin Treatment
Number of Critical Medical Assessments Related to LC-FAOD for Other Major Clinical Events | Up to 48 Weeks Prior to and 48 Weeks After the Start of Triheptanoin Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (15):
- United States (15):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Kaiser Permanente, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Duke University, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington